CLINICAL TRIAL: NCT01436838
Title: Prospective Study of Betaferon in Adherence, Coping and Nurse Support in Patients of Chinese Origin With Multiple Sclerosis
Brief Title: China Betaferon Adherence, Coping and Nurse Support Study
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15916; BF1110CN (Other: Company Internal)
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis, Chronic Progressive
Keywords: Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — All patients will be prescribed with Betaseron and be instructed on treatment by their phisicians

SUMMARY:
Non-adherence reduces treatment benefit and can bias the assessment of treatment efficacy thereby involving safety risks for the patient and influencing health cost-effectiveness. This observational study will concentrate upon the role of MS nurses in influencing adherence. This study will examine the influence of initial and subsequent periodic nurse interviews which aim to improve adherence to Betaferon® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple scelrosis (RRMS) and secondary progressive multiple sclerosis (SPMS) patients
* Having Betaferon treatment, including patients who are

  * First time using; or
  * Re-staring; or
  * Switching from other diseases modifying drugs (DMDs)

Exclusion Criteria:

* Known or newly identified contraindication for administration of Betaferon according to Summary of Product Characteristic (SmPC).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS center located in general hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adherence to Betaferon treatment: proportion of patients adhering to Betaferon treatment | at 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Ways of Coping Questionnaire (WCQ) | at 6, 12, 18 and 24 months
Hospital Anxiety and Depression Scale (HAD) | at 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China